CLINICAL TRIAL: NCT03677960
Title: Open-Label Study To Evaluate The Safety, Tolerability, And Pharmacokinetics Of Multiple Doses Of Topical Abi-1968 In Subjects With Anal High-Grade Squamous Intraepithelial Lesions (aHSIL)
Brief Title: Study of Topical ABI-1968 in Subjects With Precancerous Anal Lesions Resulting From Human Papillomavirus (HPV) Infection
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Pre-Clinical Toxicology Findings
Sponsor: Antiva Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABI-1968-202
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-04

CONDITIONS: HSIL, High-Grade Squamous Intraepithelial Lesions; Human Papilloma Virus Infection; HIV Infection; Anal Cancer; Anus Neoplasm
MeSH Terms: conditions — Squamous Intraepithelial Lesions; Papillomavirus Infections; HIV Infections; Anus Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose 1 - Multiple Ascending Dose(MAD) (Experimental): Multiple Doses of Topical ABI-1968 cream applied by the Investigator in the clinic
  Interventions: Drug: Topical ABI-1968 cream
- Dose 2 - Multiple Ascending Dose(MAD) (Experimental): Multiple Doses of Topical ABI-1968 cream applied by the Investigator in the clinic
  Interventions: Drug: Topical ABI-1968 cream
- Dose 3 - Multiple Ascending Dose(MAD) (Experimental): Multiple Doses of Topical ABI-1968 cream applied by the Investigator in the clinic
  Interventions: Drug: Topical ABI-1968 cream

INTERVENTIONS:
Drug: Topical ABI-1968 cream — Multiple doses of Topical ABI-1968 Cream administered by the Investigator in the clinic up to Day 29

SUMMARY:
This study evaluates the use of ABI-1968, a topical cream, in the treatment of anal precancerous lesions in adults with and without human immunodeficiency virus (HIV) infection

ELIGIBILITY:
Inclusion Criteria

1. Female or male subjects, at least 27 years old.
2. Confirmed diagnosis of intra-anal HSIL at least 3 months prior to screening and confirmed by histopathology (with p16 positive staining)
3. Intra-anal HSIL are visible and evaluable by HRA at the time of screening, and no lesion(s) is suspicious for invasive cancer.
4. For HIV-positive subjects, CD4 count must be at least 200/mm3 with undetectable (<50 copies/mL) viral load within the 3 months prior to enrollment. Subjects must be on a stable regimen of antiretroviral drugs for the 3 months prior to enrollment.

Exclusion Criteria:

1. Women who are pregnant, plan to become pregnant in the next 3 months, or lactating females.
2. Received topical treatment or ablative procedures for aHSIL in the 6 months prior to enrolment.
3. History of cancer involving the anogenital region, or history of other cancers that have not been fully resolved and free of symptoms in the past 5 years
4. History of genital herpes with > 3 outbreaks per year.
5. Plan to have excision or ablation of the lesion(s) within 3 months of enrolment.

Min Age: 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of ABI-1968 for the treatment of aHSIL | MAD portion is 84 days
  Number of participants with Adverse Events related to treatment

SECONDARY OUTCOMES:
Systemic exposure to ABI-1968 Topical Cream following topical application to the anal canal. | MAD portion is 84 days
  Plasma concentrations of ABI-1968 over time

OTHER OUTCOMES:
Histopathology of areas with biopsy-proven disease following multiple doses of ABI-1968 Topical Cream. | MAD portion is 84 days
  Number of subjects with complete and or partial regression of aHSIL by High Resolution Anoscopy (HRA) and histopathology

CONTACTS AND LOCATIONS:
Locations (2):
- Research Center, Chicago, Illinois, United States
- Research Center, Darlinghurst, Sydney, Australia